CLINICAL TRIAL: NCT07000110
Title: A Non-Interventional Multi-Country Post-Authorisation Safety Study (PASS) to Assess the Incidence of Serious Infections & Malignancies in Systemic Lupus Erythematosus (SLE) Patients Exposed to Anifrolumab
Brief Title: Anifrolumab Malignancy and Serious Infections Study
Acronym: SIMA
Status: Not yet recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: D3461R00046
Record Dates: First submitted 2025-05-22; First posted 2025-06-02 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Systemic Lupus Erythematosus
Keywords: malignancies, infections, anifrolumab
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Neoplasms; Infections | interventions — anifrolumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Drug: Anifrolumab — Anifrolumab prescribed per local practice
  Other Names: Saphnelo

SUMMARY:
This is an observational study, in which the main research question is to evaluate the risk of malignancies and serious infections among moderate/severe SLE patients who receive anifrolumab compared with a comparable population of moderate/severe SLE patients on standard of care who do not initiate anifrolumab.

DETAILED DESCRIPTION:
This is an observational study, in which the main research question is to evaluate the risk of malignancies and serious infections among moderate/severe SLE patients who receive anifrolumab compared with a comparable population of moderate/severe SLE patients on standard of care who do not initiate anifrolumab.

ELIGIBILITY:
Inclusion Criteria:

* First prescription of anifrolumab in the study period (no anifrolumab prescription prior to index date): date of first anifrolumab prescription will be the index date
* A minimum data availability of 12 months prior to index date
* Age ≥18 years at index date
* SLE severity: patients with moderate to severe SLE at index date
* SLE activity: patients with at least a flare (uncontrolled SLE) in the 6 months prior to index date

Exclusion Criteria:

* A diagnosis of any malignancy prior to index date
* A diagnosis of HIV/AIDS or congenital immunodeficiency prior to index date
* Organ or bone marrow transplant procedure prior to index date
* A diagnosis of serious infection in the previous 6 months

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Moderate/severe SLE patients who receive anifrolumab compared with a comparable population of moderate/severe SLE patients on standard of care (SOC) who do not initiate anifrolumab.
Sampling Method: Non-Probability Sample
Enrollment: 3506 (Estimated)
Dates: Start 2025-11-28 (Estimated); Primary Completion 2031-11-30 (Estimated); Study Completion 2031-11-30 (Estimated)

PRIMARY OUTCOMES:
Malignancies | Indexdate to November 2031
  Defined as the first coded diagnosis for hematological malignancies and solid tumors available in the data source
Serious infection | Indexdate to November 2027
  Infection leading to hospitalization, use of intravenous antimicrobials or an infection-related death
Infections leading to hospitalisation | Index date to November 2027
  Infection diagnosis as a part of a hospitalization episode, use of IV antimicrobials, or death, or infection diagnosis in primary or secondary care settings up to 7 days before hospitalization
Infection-related death | Indexdate to November 2027
  Recorded diagnosis of infection in primary or secondary care settings with record of death within the subsequent month

SECONDARY OUTCOMES:
Specific types of malignancies | Indexdate to November 2031
  Haematologic, solid and skin malignancies
Serious infection components | Indexdate to November 2027
  Infection leading to hospitalization, infection requiring treatment with IV antimicrobials and infection-related death
Serious infection types grouped as opportunistic serious infections, other serious infections, pneumonia (overall), fatal and non-fatal pneumonia (separately) | Indexdate to November 2027

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/